CLINICAL TRIAL: NCT07045246
Title: The Evaluation of the Effect of Co-enzyme Q10 on the Bone Volume of Alveolar Cleft Reconstruction (Randomized Clinical Trial)
Brief Title: Effect of Co-enzyme Q10 on the Bone Volume of Alveolar Cleft Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mennat Allah Sayed Ibrahim Ali, Demonstrator, Oral and Maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoQ10 in Cleft Reconstruction
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Coenzyme Q10; Alveolar Cleft Grafting
Keywords: alveolar cleft reconstruction
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iliac bone graft (Active Comparator): In the control group, A skin incision will be performed 1cm posterior to the anteriorsuperior iliac crest for iliac grafting. External oblique muscle and periosteum will be reflected medially to expose the anterior iliac crest. The cancellous graft will be gathered using trephine burs and surgical curettes after trap door fenestration reflection. The wound will be closed in three layers; muscle, subcutaneous, and skin. The cancellous bone will be packed to fill the alveolar defect in the control group.
  Interventions: Procedure: iliac bone graft
- CoQ10 graft (Active Comparator): the Co-enzyme Q10 will be packed into the alveolar cleft defect alone
  Interventions: Procedure: Coenzyme Q 10

INTERVENTIONS:
Procedure: Coenzyme Q 10 — Patients received Coenzyme Q 10 as a graft material in unilateral maxillary alveolar cleft
  Arms: CoQ10 graft
Procedure: iliac bone graft — iliac bone used as a graft for alveolar cleft reconstruction
  Arms: Iliac bone graft

SUMMARY:
Evaluate the effect of Co-enzyme Q10 on the bone volume in unilateral alveolar cleft repair

DETAILED DESCRIPTION:
Cleft lip or palate is the most frequent congenital abnormality, accounting for about 0.3/1000 live births in Egypt and 1/ 500-1000 live births worldwide. In 75% of patients, cleft lip and palate are accompanied by an alveolar cleft. Alveolar cleft reconstruction is needed to conserve the continuity of the arch, provide the maximum amount of bone support for the nose and permanent teeth eruption, and repair the residual oro-antral fistula. Alveolar cleft grafting is performed at various ages, but secondary grafting, performed between the ages of 9 and 12, is the most suitable and advantageous. Due to its osteogenic, osteoinductive, and osteoconductive properties, the autogenous iliac bone graft is considered the "gold standard" for alveolar cleft repair. However, the autogenous iliac bone graft is associated with a graft resorption rate of about 15-24% during the first six months. In order to resolve those complications, different substances were combined with the iliac graft, such as platelet-rich plasma (PRP), fibrin glue, or bone morphogenic protein (BMP). Nevertheless, it was demonstrated that there was no difference between iliac grafts with or without these materials. Various graft materials, such as allograft, xenograft, and synthetic bone grafts, have been utilized as an alternative to autogenous bone grafts. Allografts are expensive and associated with risks of bacterial contamination, viral transmission, and immunogenicity. Conversely, the main drawbacks of synthetic bone grafts are slow resorption and brittleness. A combination of hydroxyapatite and b-tricalcium phosphate, along with an autogenous bone graft, has been used to address these drawbacks. Co-enzyme Q10 is a lipid-soluble vitamin-like compound present in the inner membrane of the mitochondria of every cell of the body. The structure of Coenzyme Q10 consists of a benzoquinone ring and a lipophilic isoprenoid side chain with ten isoprenyl units in the case of humans, which determines its low polarity and allows its fast diffusion through mitochondrial membrane. Recently, Coenzyme Q10 has gained attention for its therapeutic application for several disorders including cardiovascular diseases, inflammation, human fertility, and diabetes mellitus. Co-enzyme Q10 provides membrane stabilizing properties and acts as an antioxidant with cell-protective effect which acts as an inhibitor of RANKLinduced osteoclast differentiation and enhancer of bone-forming osteoblast differentiation. Co-enzyme Q10 leads to a decreased TRAP+ MNCs formation, as well as dose-dependent down regulation of gene expressions, NFATc1, TRAP, and OSCAR, for osteoclast differentiation. Co-enzyme Q10 in high concentrations (over 10 µM) disturbed the production of ROS and attenuates the H2O2-induced early signaling activities including p38, IκBα, and JNK signaling pathways. Additionally, Co-enzyme Q10 furthered the induction of osteoblastogenic gene markers and also promoted matrix mineralization by enhancing bone nodule formation. Co-enzyme Q10 treatment is safe, even at the highest doses. Most clinical trials have not reported significant adverse effects that necessitated stopping therapy. It undergoes biotransformation in the liver and is eliminated primarily via the biliary tract; therefore it can accumulate in patients with hepatic impairment or biliary obstruction. Many studies used Co-enzyme Q10 in bone augmentation and socket preservation. The use of Co-enzyme Q10 enhances the bone quality and decreases the rate of bone resorption. No study has investigated the effect of the Co-enzyme Q10 in the reconstruction of the alveolar cleft, despite its role in bone healing. Consequently, the present study targeted to assess the significance of Co-enzyme Q10 on the quality and quantity of bone formation in unilateral alveolar cleft repair

ELIGIBILITY:
Inclusion Criteria:

* age ranged between 10-14 years, with good oral hygiene and general good health

Exclusion Criteria:

* patients with syndromes associated with an alveolar cleft, local pathosis at the maxilla that may interfere with surgery, previous grafting attempts, or cleft palate fistulae

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
bone volume | 6 months postoperative
  V= (A1xT) + (A2 xT) + …….+ (An xT) where: V= volume A= area T= thickness of the axial C.T slice N=number of Slices

SECONDARY OUTCOMES:
bone density | 6 months postoperative
  the average bone density will be measured from the CBCT
bone formation ratio | 6 months postoperative
  BF% = (formed volume/alveolar defect) ×100%

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Faculty of Dentistry, Al Fayyum, Egypt

REFERENCES:
- [Background] Shabaan AA, Salahuddin A, Aboulmagd I, Ragab R, Salah KA, Rashid A, Ayad HM, El Aty Ahmed WA, Refahee SM. Alveolar cleft reconstruction using bone marrow aspirate concentrate and iliac cancellous bone: A 12-month randomized clinical study. Clin Oral Investig. 2023 Nov;27(11):6667-6675. doi: 10.1007/s00784-023-05276-9. Epub 2023 Oct 5. PMID 37794139
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4176102/